CLINICAL TRIAL: NCT00890760
Title: Assessment of Protection Against Malaria by Sporozoite Challenge of Healthy Adults Vaccinated With AdCh63 ME-TRAP and MVA ME-TRAP
Brief Title: A Study to Assess the Effectiveness of a New Malaria Vaccine Candidate by Infecting Vaccinated Volunteers With Malaria Parasites
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Professor Adrian VS Hill, Centre for Clinical Vaccinology and Tropical Medicine University of Oxford
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MAL 034
Record Dates: First submitted 2009-04-29; First posted 2009-04-30 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-11

CONDITIONS: Malaria
Keywords: Malaria; Vaccine
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- Group 1 (Experimental): AdCh63 ME-TRAP prime followed by MVA ME-TRAP boost 8 weeks later and challenged by sporozoite 3 weeks after boost
  Interventions: Biological: AdCh63 ME-TRAP; Biological: MVA ME-TRAP; Other: Sporozoite challenge
- Group 2 (Experimental): AdCh63 ME-TRAP alone followed by sporozoite challenge 3 weeks later
  Interventions: Biological: AdCh63 ME-TRAP; Other: Sporozoite challenge
- Group 3 (Experimental): Non-vaccinated Control for Groups 1 and 2 challenged with sporozoite
  Interventions: Other: Sporozoite challenge
- Group 4 (Experimental): AdCh63 ME-TRAP prime followed by MVA ME-TRAP boost 8 weeks later and challenged by sporozoite 11 weeks after boost
  Interventions: Biological: AdCh63 ME-TRAP; Biological: MVA ME-TRAP; Other: Sporozoite challenge
- Group 5 (Experimental): AdCh63 ME-TRAP prime followed by MVA ME-TRAP boost 8 weeks later and challenged by sporozoite 3 weeks after boost
  Interventions: Biological: AdCh63 ME-TRAP; Biological: MVA ME-TRAP; Other: Sporozoite challenge
- Group 6 (Experimental): Protected volunteers from Group 1 re-challenged with sporozoite after 6 months
  Interventions: Biological: AdCh63 ME-TRAP; Other: Sporozoite challenge
- Group 7 (Experimental): Non vaccinated control for Groups 4-6, 8-10 challenged with sporozoite
  Interventions: Other: Sporozoite challenge
- Group 8 (Experimental): 3 vaccinations of mixture formulation AdCh63 ME-TRAP and MVA ME-TRAP give at 8 weeks interval each followed by sporozoite challenge 3 weeks after last vaccination
  Interventions: Other: Sporozoite challenge; Biological: Mixture of AdCh63 ME-TRAP and MVA ME-TRAP intramuscularly
- Group 9 (Experimental): 2 vaccinations of mixture formulation AdCh63 ME-TRAP and MVA ME-TRAP give at 8 weeks interval followed by sporozoite challenge 3 weeks after last vaccination
  Interventions: Other: Sporozoite challenge; Biological: Mixture of AdCh63 ME-TRAP and MVA ME-TRAP intramuscularly
- Group 10 (Experimental): 3 vaccinations of mixture formulation AdCh63 ME-TRAP and MVA ME-TRAP give at 4 weeks interval each followed by sporozoite challenge 3 weeks after last vaccination
  Interventions: Other: Sporozoite challenge; Biological: Mixture of AdCh63 ME-TRAP and MVA ME-TRAP intramuscularly

INTERVENTIONS:
Biological: AdCh63 ME-TRAP — 5 x 10*10 vp IM
  Arms: Group 1; Group 2; Group 4; Group 5; Group 6
Biological: MVA ME-TRAP — 2 x 10*8 pfu ID
  Arms: Group 1; Group 4; Group 5
Other: Sporozoite challenge — Infected mosquito bite
Biological: Mixture of AdCh63 ME-TRAP and MVA ME-TRAP intramuscularly — AdCh63 ME-TRAP 5 x 10*10 vp MVA ME-TRAP 2 x 10*8 pfu
  Arms: Group 10; Group 8; Group 9

SUMMARY:
Malaria affects around 515 million people each year, about a million of whom die from the disease. It is a major problem for those who live in affected areas as well as for travellers to affected areas. There is a great need for a safe, effective malaria vaccine. The purpose of this study is to test 2 new vaccination regimes that include a new malaria vaccine candidate, for their ability to prevent malaria infection.

The vaccines are different types of virus which contain genetic information (DNA) from the malaria parasite. This genetic material is named ME-TRAP. The aim is to use these viruses to help the body make an immune response against the malaria parasite. Both viruses are inactivated so that they are unable to multiply within the body.

The first vaccine virus is a weakened version of a common cold virus. Such adenoviruses occur in many strain types and commonly infect chimpanzees as well as people and this vaccine uses a strain originally derived from a chimpanzee. The vaccine is called AdCh63 ME-TRAP.

The other virus is Modified Vaccinia Ankara Virus, (MVA), which is a safer form of the vaccine virus previously widely used for smallpox vaccination. The vaccine is called MVA ME-TRAP.

This study will enable the investigators to assess:

1. The ability of different vaccine combinations to prevent malaria infection
2. The safety of the vaccine combinations in healthy volunteers
3. The response of the human immune system to the vaccines

ELIGIBILITY:
Inclusion Criteria:

* Able and willing (in the Investigator's opinion) to comply with all study requirements
* Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner
* For females only: willingness to practise effective contraception throughout the study
* Agreement to refrain from blood donation during the course of the study
* Written informed consent

Exclusion Criteria:

* Participation in another research study involving an investigational product in the 30 days preceding enrolment, or planned use during the study period.
* Prior receipt of an investigational malaria vaccine encoding ME-TRAP or any other investigational vaccine likely to impact on interpretation of the trial data
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
* Pregnancy, lactation or intention to become pregnant during the study
* Contraindication to both anti-malarial drugs (Riamet® and chloroquine)

  o concomitant use with other drugs known to cause QT-interval prolongation, ( e.g. macrolides, quinolones, amiodarone etc)
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, e.g. egg products, Kathon.
* History of clinically significant contact dermatitis
* Any history of anaphylaxis in reaction to vaccination
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
* History of serious psychiatric condition
* Any other serious chronic illness requiring hospital specialist supervision
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week
* Suspected or known injecting drug abuse
* Seropositive for hepatitis B surface antigen (HBsAg)
* Seropositive for hepatitis C virus (antibodies to HCV)
* Seropositive for simian adenovirus 63 (antibodies to AdCh63) at a titre > 1: 200 ( EXCEPT CONTROL VOLUNTEERS)
* Any other significant disease, disorder or finding, which, in the opinion of the Investigator, may either put the volunteer at risk because of participation in the study, or may influence the result of the study, or the volunteer's ability to participate in the study.
* History of clinical P. falciparum malaria
* Travel to a malaria endemic region during the study period or within the previous six months
* Any clinically significant abnormal finding on screening biochemistry or haematology blood tests or urinalysis
* Any other finding which in the opinion of the investigators would significantly increase the risk of having an adverse outcome from participating in the protocol or impair interpretation of the study data.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2009-03; Primary Completion 2010-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Vaccine prevention (partial or complete) of malaria infection by sporozoite challenge | Approxiamately 5-16 months following last intervention

SECONDARY OUTCOMES:
Safety of vaccine | Approxiamately 5-16 months following last intervention

CONTACTS AND LOCATIONS:
Overall Officials: Adrian VS Hill, D.Phil, FRCP, Principal Investigator — University of Oxford
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine, University of Oxford, Oxford, Headington, United Kingdom

REFERENCES:
- [Derived] Ewer KJ, O'Hara GA, Duncan CJ, Collins KA, Sheehy SH, Reyes-Sandoval A, Goodman AL, Edwards NJ, Elias SC, Halstead FD, Longley RJ, Rowland R, Poulton ID, Draper SJ, Blagborough AM, Berrie E, Moyle S, Williams N, Siani L, Folgori A, Colloca S, Sinden RE, Lawrie AM, Cortese R, Gilbert SC, Nicosia A, Hill AV. Protective CD8+ T-cell immunity to human malaria induced by chimpanzee adenovirus-MVA immunisation. Nat Commun. 2013;4:2836. doi: 10.1038/ncomms3836. PMID 24284865